CLINICAL TRIAL: NCT06943586
Title: Pharmacogenomics in Stroke: Feasibility of CYP2C19 Testing in Patients With Minor Stroke or High Risk TIA (CYP2C19 and Stroke)
Brief Title: Pharmacogenomics in Stroke: Feasibility of CYP2C19 Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ekaterina Bakradze, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-300013920; MULTIPI8165 (Other Grant/Funding Number: University of Alabama at Birmingham)
Record Dates: First submitted 2025-04-03; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Transient Ischemic Attack (TIA)
Keywords: Personalized medicine; CYP2C19; minor stroke; Transient Ischemic Attack; TIA
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Intervention Model Description: Participants will undergo collection of buccal swabs for CYP2C19 testing and be randomized (depending on CYP2C19 strata- normal vs. loss-of-function (LOF)* CYP2C19 allele) to their assigned study medications (aspirin and clopidogrel vs aspirin and ticagrelor).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CYP2C19 strata-normal (Active Comparator): Participants undergo buccal swab for genetic testing to determine potential medication response to standard of care (SOC) medications. Upon result, participants are randomized (1:1) to aspirin and clopidogrel vs aspirin and ticagrelor (all SOC for this stroke population). Doses are aspirin either 81mg or loading dose 325mg, clopidogrel either 75mg or loading dose 300mg, ticagrelor either 90mg or loading dose 180mg. Loading doses are given once for aspirin, clopidogrel or ticagrelor; aspirin 81mg is taken once a day for the duration of the study; clopidogrel 75mg is once a day for 21 days only, ticagrelor 90mg is twice daily for 21 days. Participants will only receive loading dose of aspirin if not already taken at home. CYP2C19 results only affect decision regarding clopidogrel and ticagrelor but not aspirin. Aspirin is not affected by CYP2C19 mutation and will be given immediately without waiting for CYP2C19 results.
  Interventions: Genetic: CYP2C19 Genotype Guided DAPT (dual antiplatelet therapy)
- loss-of-function CYP2C19 allele (Active Comparator): Participants undergo buccal swab for genetic testing to determine potential medication response to standard of care (SOC) medications. Upon result, participants are randomized (1:1) to aspirin and clopidogrel vs aspirin and ticagrelor (all SOC for this stroke population). Doses are aspirin either 81mg or loading dose 325mg, clopidogrel either 75mg or loading dose 300mg, ticagrelor either 90mg or loading dose 180mg. Loading doses are given once for aspirin, clopidogrel or ticagrelor; aspirin 81mg is taken once a day for the duration of the study; clopidogrel 75mg is once a day for 21 days only, ticagrelor 90mg is twice daily for 21 days. Participants will only receive loading dose of aspirin if not already taken at home. CYP2C19 results only affect decision regarding clopidogrel and ticagrelor but not aspirin. Aspirin is not affected by CYP2C19 mutation and will be given immediately without waiting for CYP2C19 results.
  Interventions: Genetic: CYP2C19 Genotype Guided DAPT (dual antiplatelet therapy)

INTERVENTIONS:
Genetic: CYP2C19 Genotype Guided DAPT (dual antiplatelet therapy) — CYP2C19 is a gene that encodes an enzyme responsible for metabolizing several medications, including the antiplatelet drugs.
  Other Names: genotype guided antiplatelet treatment

SUMMARY:
The purpose of this research study is to explore whether genetic testing can offer a personalized and timely approach to assist physicians in making more informed medication decisions for stroke or high-risk transient ischemic attack (TIA) patients during their hospital stay.

DETAILED DESCRIPTION:
This is a pilot clinical trial for feasibility

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-89 years of age
* admitted to University of Alabama at Birmingham (UAB) main hospital with symptoms or signs of minor ischemic stroke, or high risk TIA
* eligible to receive dual antiplatelet load (presented to the hospital within 66 hours of last known well)

Exclusion Criteria:

* diagnosis of atrial fibrillation, valvular heart disease, index stroke due to known hypercoagulability (subset of other determined etiology) or large vessel disease (culprit vessel stenosis of ≥50%)
* prescribed anticoagulation prior to stroke
* treated with intravenous thrombolysis
* treated with mechanical thrombectomy
* missing NIH Stroke Scale score

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Stroke participant feasibility of return of CYP2C19 genetic testing results | 6 hours from buccal swab collection
  This outcome is to determine the feasibility of receiving CYP2C19 genetic testing results (strata-normal vs. loss-of-function allele) on minor ischemic stroke and high risk TIA inpatients within a 6-hour window to determine drug metabolization for antiplatelet effect to guide standard of care treatment. Inpatients that have been admitted to the hospital, within 66 hours of last known well time, will have buccal swabs collected during hospitalization for the CYP2C19 genetic testing. Results must be received within 6 hours to effectively randomize subjects.

SECONDARY OUTCOMES:
Recurrent stroke, TIA, major bleeding and Modified Rankin Scale at ~90days | 90 days following stroke
  Participants will undergo a visit approximately 90 days following stroke to assess for any new stroke like symptoms and recovery in daily activities via the modified Rankin scale (mRS) Score. The mRS is a widely used tool to assess functional outcome after a stroke or other neurological events, ranging from 0 (no symptoms) to 6 (dead), with higher scores indicating greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Bakradze, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot clinical trial for feasibility

REFERENCES:
- [Background] Nordeen JD, Patel AV, Darracott RM, Johns GS, Taussky P, Tawk RG, Miller DA, Freeman WD, Hanel RA. Clopidogrel Resistance by P2Y12 Platelet Function Testing in Patients Undergoing Neuroendovascular Procedures: Incidence of Ischemic and Hemorrhagic Complications. J Vasc Interv Neurol. 2013 Jun;6(1):26-34. PMID 23826440
- [Background] Meschia JF, Walton RL, Farrugia LP, Ross OA, Elm JJ, Farrant M, Meurer WJ, Lindblad AS, Barsan W, Ching M, Gentile N, Ross M, Nahab F, Easton JD, Kim AS, Zurita KG, Cucchiara B, Johnston SC. Efficacy of Clopidogrel for Prevention of Stroke Based on CYP2C19 Allele Status in the POINT Trial. Stroke. 2020 Jul;51(7):2058-2065. doi: 10.1161/STROKEAHA.119.028713. Epub 2020 Jun 17. PMID 32568642
- [Background] Wang Y, Meng X, Wang A, Xie X, Pan Y, Johnston SC, Li H, Bath PM, Dong Q, Xu A, Jing J, Lin J, Niu S, Wang Y, Zhao X, Li Z, Jiang Y, Li W, Liu L, Xu J, Chang L, Wang L, Zhuang X, Zhao J, Feng Y, Man H, Li G, Wang B; CHANCE-2 Investigators. Ticagrelor versus Clopidogrel in CYP2C19 Loss-of-Function Carriers with Stroke or TIA. N Engl J Med. 2021 Dec 30;385(27):2520-2530. doi: 10.1056/NEJMoa2111749. Epub 2021 Oct 28. PMID 34708996
- [Background] Pereira NL, Cresci S, Angiolillo DJ, Batchelor W, Capers Q 4th, Cavallari LH, Leifer D, Luzum JA, Roden DM, Stellos K, Turrise SL, Tuteja S; American Heart Association Professional/Public Education and Publications Committee of the Council on Genomic and Precision Medicine; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Peripheral Vascular Disease; and Stroke Council. CYP2C19 Genetic Testing for Oral P2Y12 Inhibitor Therapy: A Scientific Statement From the American Heart Association. Circulation. 2024 Aug 6;150(6):e129-e150. doi: 10.1161/CIR.0000000000001257. Epub 2024 Jun 20. PMID 38899464
- [Background] Prevention: Cfdca. Centers for disease control and prevention: Stroke. Accessed May 18, 2023